CLINICAL TRIAL: NCT04134715
Title: A PHASE 1, RANDOMIZED, OPEN LABEL, FIXED SEQUENCE STUDY TO ESTIMATE THE EFFECT OF PF-06826647 ON THE PHARMACOKINETICS OF ORAL CONTRACEPTIVE STEROIDS AND TO ESTIMATE THE EFFECT OF ORAL CONTRACEPTIVE STEROIDS ON PHARMACOKINETICS OF PF-06826647 IN HEALTHY FEMALE PARTICIPANTS
Brief Title: A Drug Drug Interaction Study Between PF-06826647 And Oral Contraceptive Steroids In Healthy Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: C2501005
Record Dates: First submitted 2019-09-04; First posted 2019-10-22 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Healthy
Keywords: Oral contraceptive; Drug-Drug Interaction (DDI); PF-06826647
MeSH Terms: interventions — ropsacitinib; Contraceptives, Oral

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-06826647 alone then OC alone then OC+PF-06826647 (Experimental): In Period 1 (Period 1 is 2 days), participants will receive a single dose of PF-06826647 600 mg on Day 1. Period 2 (Period 2 is 14 days) will immediately follow Period 1 without any washout. In Period 2, the participants will receive OC in the form of 1 PORTIA (30 µg EE and 150 µg LN) or equivalent tablet, orally starting from Period 2 Day 1 until Period 3-Day 16 (Period 3 is 17 Days). Period 3 will immediately follow Period 2 with no washout. In Period 3 on Day 1, the participants will receive a single dose of PF-06826647 600 mg. On Day 2 in Period 3, PF-06826647 will not be dosed. From Day 3, the participants will receive PF-06826647 600 mg QD for 14 days followed by OC in the form of 1 PORTIA (EE and LN) or equivalent tablet.
  Interventions: Drug: PF-06826647; Drug: Oral Contraceptive (OC)

INTERVENTIONS:
Drug: PF-06826647 — 100 mg tablet
Drug: Oral Contraceptive (OC) — OC in the form of 1 PORTIA (30 µg EE and 150 µg LN) or equivalent tablet

SUMMARY:
This is a Phase 1, fixed sequence, multiple dose, open label study of the effect of PF-06826647 on oral contraceptive (OC) pharmacokinetics (PK) and vice versa in healthy female participants. A total of approximately 15 healthy female participants will be enrolled and dosed to achieve at least 12 participants completing the study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy female participants of non-childbearing potential must be 18 to 60 years of age, inclusive
* 2. Female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, including blood pressure (BP) and pulse rate measurement, laboratory tests, and 12 lead ECG
* 3. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures
* 4. Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb)

Exclusion Criteria:

* 1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* 2. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* 3. History of venous and arterial thrombosis (ie, deep venous thrombosis, pulmonary embolism) or hereditary clotting disorders (in first degree immediate relatives).
* 4. History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCVAb). Hepatitis B vaccination is allowed.
* 5. Any current evidence of untreated active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB).
* 6. Participants who use tobacco or nicotine containing products.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women of non-child bearing potential
Enrollment: 15 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Profile From Time Zero To End of Dosing Interval (AUGtau) of Ethinyl Estradiol (EE) | Day 14 in Period 2 (Period 2 is 14 days) and Day 16 in Period 3 (Period 3 is 17 days)
  Area under the plasma concentration time profile from time 0 to end of dosing interval (AUCtau), where dosing interval is 24 hours.
Area Under the Plasma Concentration-Time Profile From Time Zero To End of Dosing Interval (AUGtau) of Levonorgestrel (LN) | Day 14 in Period 2 (Period 2 is 14 days) and Day 16 in Period 3 (Period 3 is 17 days)
  Area under the plasma concentration time profile from time 0 to end of dosing interval (AUCtau), where dosing interval is 24 hours.
Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of PF-06826647 | Day 1 in Period 1 (Period 1 is 2 days) and Period 3 (Period 3 is 17 days)
  AUCinf is calculated by AUClast + (Clast*/kel), where AUClast is the area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration, Clast* is the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis, and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Maximum Plasma Concentration (Cmax) of PF-06826647 | Day 1 in Period 1 (Period 1 is 2 days) and Period 3 (Period 3 is 17 days)
  Cmax will be observed directly from data.

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Baseline in Period 1 (Period 1 is 2 days) to Day 17 in Period 3 (Period 3 is 17 days)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A serious adverse event (SAE) is defined as any untoward medical occurrence at any dose that results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; results in congenital anomaly/birth defect. AEs include both SAEs and AEs. TEAEs are AEs that occur following the start of treatment or AEs increasing in severity during treatment.
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline in Period 1 (Period 1 is 2 days) to Day 17 in Period 3 (Period 3 is 17 days)
  Vital signs evaluation includes: supine systolic and diastolic blood pressure (BP), and pulse rate.
Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)-Hematology | Baseline in Period 1 (Period 1 is 2 days) to Day 17 in Period 3 (Period 3 is 17 days)
  Hematology evaluation includes: hemoglobin, hematocrit, red blood cell (RBC) count, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), platelets, white blood cell count (WBC), neutrophils, eosinophils, monocytes, basophils, lymphocytes and reticulocytes.
Number of Participants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)-Clinical Chemistry | Baseline in Period 1 (Period 1 is 2 days) to Day 17 in Period 3 (Period 3 is 17 days)
  Clinical chemistry evaluation includes: blood urea nitrogen, creatinine, fasting glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase, alanine aminotransferase, bilirubin, alkaline phosphatase, urate, albumin, protein, creatinine kinase
Number of Paticipants With Laboratory Test Abnormalities (Without Regard to Baseline Abnormality)-Urinalysis | Baseline in Period 1 (Period 1 is 2 days) to Day 17 in Period 3 (Period 3 is 17 days)
  Urinalysis evaluation includes: qual urine glucose, qual protein, qual blood, ketones, nitrites, leukocyte esterase, urobilinogen, urine bilirubin, urine leukocytes.
Number of Participants with Clinically Significant Change From Baseline in Electrocardiogram (ECG) Findings | Baseline (Period 1 Day 1), Day 1 (Period 1 and Period 2) up to Day 17 (Period 3)
  Criteria for clinically significant changes in ECG (12-lead) are defined as: a postdose QTc interval increase by ≥30 msec from the baseline and is >450 msec; or an absolute QTc value is ≥500 msec for any scheduled ECG

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Quotient Sciences Screening Office, Coral Gables, Florida
  - Quotient Sciences-Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2501005